CLINICAL TRIAL: NCT04414345
Title: HEALEY ALS Platform Trial - Regimen C CNM-Au8
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Merit E. Cudkowicz, MD (Other)
Collaborators: Clene Nanomedicine (Industry)
Responsible Party: Sponsor-Investigator, Merit E. Cudkowicz, MD, Chief, Neurology Department, Massachusetts General Hospital
Organization: Massachusetts General Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2019P003518C
Record Dates: First submitted 2020-06-01; First posted 2020-06-04 (Actual); Results first posted 2023-07-25 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2023-06

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: ALS; Placebo-Controlled; Double-Blind; Regimen-Specific Appendix; Lou Gehrig's Disease; CNM-Au8; Clene Nanomedicine
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CNM-Au8 (Experimental): Drug: CNM-Au8
  Administration: Oral
  Dosage: 30 mg or 60 mg daily
  Interventions: Drug: CNM-Au8
- Matching Placebo (Placebo Comparator): Administration: Oral
  Dosage: 2 bottles daily
  Interventions: Drug: Matching Placebo

INTERVENTIONS:
Drug: CNM-Au8 — Drug: CNM-Au8
  Administration: Oral
  Dosage: 30 mg or 60 mg daily
  Arms: CNM-Au8
Drug: Matching Placebo — Drug: Matching Placebo
  Administration: Oral
  Dosage: 2 bottles daily
  Arms: Matching Placebo

SUMMARY:
The HEALEY ALS Platform Trial is a perpetual multi-center, multi-regimen clinical trial evaluating the safety and efficacy of investigational products for the treatment of ALS.

Regimen C will evaluate the safety and efficacy of a single study drug, CNM-Au8, in participants with ALS.

DETAILED DESCRIPTION:
The HEALEY ALS Platform Trial is a perpetual multi-center, multi-regimen clinical trial evaluating the safety and efficacy of investigational products for the treatment of ALS. This trial is designed as a perpetual platform trial. This means that there is a single Master Protocol dictating the conduct of the trial. The HEALEY ALS Platform Trial Master Protocol is registered as NCT04297683.

Once a participant enrolls into the Master Protocol and meets all eligibility criteria, the participant will be eligible to be randomized into any currently enrolling regimen. All participants will have an equal chance of being randomized to any currently enrolling regimen.

If a participant is randomized to Regimen C - CNM-Au8, the participant will complete a screening visit to assess additional Regimen C eligibility criteria. Once Regimen C eligibility criteria are confirmed, participants will complete a baseline assessment and be randomized in a 3:1 ratio to either active CNM-Au8 or matching placebo.

Regimen C will enroll by invitation, as participants may not choose to enroll in Regimen C. Participants must first enroll into the Master Protocol and be eligible to participate in the Master Protocol before being able to be randomly assigned to Regimen C.

For a list of enrolling sites, please see the HEALEY ALS Platform Trial Master Protocol under NCT04297683.

ELIGIBILITY:
Inclusion Criteria:

* No additional inclusion criteria beyond the inclusion criteria specified in the Master Protocol (NCT NCT04297683).

Exclusion Criteria:

* The following exclusion criterion is in addition to the exclusion criteria specified in the Master Protocol (NCT NCT04297683).

  1. History of allergy to gold, gold salts, or colloidal gold preparations.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 161 (Actual)
Dates: Start 2020-07-30 (Actual); Primary Completion 2022-04-13 (Actual); Study Completion 2023-03-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Merit Cudkowicz, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Healey Center for ALS at Mass General, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Writing Committee for the HEALEY ALS Platform Trial; Berry JD, Maragakis NJ, Macklin EA, Chibnik LB, Quintana M, Saville BR, Detry MA, Vestrucci M, Marion J, McGlothlin A, Stommel EW, Chase M, Pothier L, Harkey BA, Yu H, Sherman A, Shefner J, Hall M, Kittle G, Babu S, Andrews J, D'Agostino D, Tustison E, Scirocco E, Giacomelli E, Alameda G, Locatelli E, Ho D, Quick A, Ajroud-Driss S, Katz J, Heitzman D, Appel SH, Shroff S, Felice KJ, Simmons Z, Miller T, Olney N, Weiss MD, Goutman SA, Fernandes JA Jr, Jawdat O, Owegi MA, Foster L, Vu T, Ilieva H, Newman DS, Arcila-Londono X, Jackson C, Ladha S, Heiman-Patterson T, Caress J, Swenson A, Peltier A, Lewis R, Fee D, Elliott M, Bedlack R, Kasarskis EJ, Elman L, Rosenfeld J, Walk D, McIlduff CE, Twydell P, Young E, Johnson K, Rezania K, Goyal NA, Cohen JA, Benatar M, Jones V, Glass J, Shah J, Beydoun SR, Wymer JP, Zilliox L, Nayar S, Pattee GL, Martinez-Thompson J, Rynders A, Evan J, Evan J, Hartford A, Sepassi M, Ho KS, Glanzman R, Greenberg B, Hotchkin MT, Paganoni S, Cudkowicz ME; HEALEY ALS Platform Trial Study Group. CNM-Au8 in Amyotrophic Lateral Sclerosis: The HEALEY ALS Platform Trial. JAMA. 2025 Feb 17;333(13):1138-49. doi: 10.1001/jama.2024.27643. Online ahead of print. PMID 40067821

RESULTS

PARTICIPANT FLOW:
Groups:
- CNM-Au8: Drug: CNM-Au8
  Administration: Oral
  Dosage: 30 mg or 60 mg daily
  CNM-Au8: Drug: CNM-Au8
  Administration: Oral
  Dosage: 30 mg or 60 mg daily
- Matching Placebo: Administration: Oral
  Dosage: 2 bottles daily
  Matching Placebo: Drug: Matching Placebo
  Administration: Oral
  Dosage: 2 bottles daily
Period: Overall Study
Arm/Group | CNM-Au8 | Matching Placebo
Started | 120 | 41
Completed | 110 | 35
Not Completed | 10 | 6

BASELINE CHARACTERISTICS:
Population: Baseline Analysis Population includes only placebo participants from the Regimen C Efficacy Regimen Only (ERO) sample; shared placebo participants from other regimens are not included in the Baseline Analysis Population.
Groups:
- Total: Total of all reporting groups
Arm/Group | CNM-Au8 | Matching Placebo | Total
Number analyzed (Participants) | 120 | 41 | 161
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.2 (9.99) | 57.0 (11.72) | 57.9 (10.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49 | 12 | 61
  Male | 71 | 29 | 100
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 3 | 6
  Not Hispanic or Latino | 116 | 38 | 154
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 2 | 2
  White | 120 | 38 | 158
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
El Escorial Diagnosis [Count of Participants; unit: Participants]
  Clinically Definite ALS | 58 | 14 | 72
  Clinically Probable ALS | 43 | 10 | 53
  Clinically Probable ALS - Laboratory Supported | 16 | 16 | 32
  Clinically Possible ALS | 3 | 1 | 4
Time Since Symptom onset at Baseline [Mean (Standard Deviation); unit: months] | 22.7 (8.64) | 21.9 (8.49) | 22.5 (8.58)
Delay in ALS Symptom Onset and Diagnosis [Mean (Standard Deviation); unit: months] | 10.5 (5.92) | 10.0 (5.64) | 10.3 (5.84)
ALS Onset Location [Count of Participants; unit: Participants]
  Bulbar | 18 | 6 | 24
  Limb | 102 | 35 | 137
Baseline Edaravone Use [Count of Participants; unit: Participants]
  No | 92 | 31 | 123
  Yes | 28 | 10 | 38
Baseline Riluzole Use [Count of Participants; unit: Participants]
  No | 26 | 9 | 35
  Yes | 94 | 32 | 126
ALSFRS-R Total Score [Mean (Standard Deviation); unit: scores on a scale] — The ALS Functional Rating Scare-Revised (ALSFRS-R) measures 12 aspects of physical function. Each of the 12 questions assessing distinct functional ability is scored from4(normal) to 0 (no ability), with a maximum total score of 48 and a minimum total score of 0. Patients with higher scores have more physical function.
  scores on a scale | 34.3 (6.56) | 36.1 (5.91) | 34.7 (6.43)
Change in ALSFRS-R prior to Baseline [Mean (Standard Deviation); unit: points per month] — The ALS Functional Rating Scare-Revised (ALSFRS-R) measures 12 aspects of physical function. Each of the 12 questions assessing distinct functional ability is scored from4(normal) to 0 (no ability), with a maximum total score of 48 and a minimum total score of 0.
  Baseline decline in ALSFRS-R was calculated as 48minus the ALSFRS-R total score at Baseline. The difference between 48 and ALSFRS-R total score at Baseline is divided by the number of months between onset of weakness due to ALS and the date of Baseline.
  A higher number indicates greater decline.
  points per month | 0.72 (0.535) | 0.60 (0.353) | 0.69 (0.497)
SVC [Mean (Standard Deviation); unit: percent predicted] — Population: Number analyzed in row differs from overall number due to missing data.
  percent predicted
    number analyzed (Participants) | 116 | 40 | 156
    (all) | 75.2 (16.08) | 76.1 (16.79) | 75.4 (16.22)
Kings Stage [Count of Participants; unit: Participants] — The King's ALS Clinical Staging System is a 4-level ordinal scale with the first three levels indicating the number (1, 2, or 3) of distinct central nervous system regions (bulbar, upper limb, and lower limb) with neuromuscular dysfunction. Level 4a indicates nutritional failure and level 4b indicates respiratory failure. Higher scores indicate a worse disease state.
  Participants
    1 Region with Neuromuscular Dysfunction | 13 | 9 | 22
    2 Regions with Neuromuscular Dysfunction | 36 | 11 | 47
    3 Regions with Neuromuscular Dysfunction | 41 | 7 | 48
    4a/b Nutritional/Respiratory Failure | 1 | 0 | 1
    4b Respiratory Failure | 29 | 14 | 43
Weight [Mean (Standard Deviation); unit: kg] | 79.6 (16.74) | 87.1 (20.38) | 81.5 (17.97)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 27.0 (5.07) | 28.4 (5.47) | 27.4 (5.20)
Serum Creatinine Concentration [Mean (Standard Deviation); unit: mg/dL] | 0.7 (0.17) | 0.7 (0.20) | 0.7 (0.18)
Neurofilament Light (NfL) Protein in Serum [Mean (Standard Deviation); unit: ng/L] — Population: Number analyzed in row differs from overall number due to missing data.
  ng/L
    number analyzed (Participants) | 117 | 39 | 156
    (all) | 91.6 (58.04) | 85.3 (71.63) | 90.0 (61.53)

OUTCOME MEASURES:

1. Primary Outcome: Disease Progression as Assessed by the ALSFRS-R Total Score
Description: Change in disease severity as measured by the ALS Functional Rating Scale-Revised (ALSFRS-R) total score using a Bayesian repeated measures model that accounts for loss to follow-up due to mortality. Each type of function is scored from 4 (normal) to 0 (no ability), with a maximum total score of 48 and a minimum total score of 0. Patients with higher scores have more physical function.
Time Frame: Baseline to 24 Weeks
Population: Outcome measure data was analyzed using the Full Analysis Set, which included shared placebo from other regimens, as pre-specified in the Regimen Statistical Analysis Plan. Regimen A Zilucoplan (NCT04436497), Regimen B Verdiperstat (NCT04436510), and Regimen D Pridopidine (NCT04615923) contributed placebo participants into the shared placebo cohort used for analysis.
Measure: Mean (Standard Deviation); unit: ALSFRS-R total score points per month
Arm/Group | CNM-Au8 | Matching Placebo
Number analyzed (Participants) | 120 | 164
ALSFRS-R total score points per month | -1.01 (0.075) | -1.03 (0.072)
Statistical Analysis 1: Comparison: CNM-Au8 vs Matching Placebo; Test type: Superiority; Bayesian shared-parameter model — Posterior probability that the disease rate ratio (DRR) is less than 1 (i.e. CNM-Au8 slowed progression) was 0.59059. NOTE: p-value is not provided for Bayesian model; A Bayesian shared-parameter model of change in disease severity as measured by ALSFRS-R total score and mortality; Disease Rate Ratio = 0.98, 95% CI 2-sided [0.797 to 1.188], Standard Deviation 0.100 — DDR <1 imply slowing of disease progression by CNM-Au8 relative to placebo. Note: reported "Confidence Interval" is actually a Bayesian credible interval; The DRR parameter for active treatment represents the relative change to the rate of decline of ALSFRS-R and the rate of mortality of treated participant relative to a placebo participant. The estimated DRR can also be interpreted as the average rate of decline in function and mortality. The model includes covariates for baseline use of edaravone, baseline use of riluzole, months since onset of symptoms, and pre-baseline slope of ALSFRS-R, and random effects for regimen and participant-specific slopes

2. Primary Outcome: Mortality Event Rate
Description: Mortality is defined as death or death equivalent. A participant is determined to meet the criteria of death equivalent if permanent assisted ventilation (PAV) is used for more than 22 hours per day for more than seven days in a row. The rate of mortality was estimated from a Bayesian shared-parametric model that assumed exponentially distributed survival times.
Time Frame: Baseline to 24 Weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: events per month
Arm/Group | CNM-Au8 | Matching Placebo
Number analyzed (Participants) | 120 | 164
events per month | 0.006 (0.002) | 0.007 (0.002)

3. Secondary Outcome: Respiratory Function
Description: Change in respiratory function as assessed by slow vital capacity (SVC).
Time Frame: Baseline to 24 Weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | CNM-Au8 | Matching Placebo
Number analyzed (Participants) | 120 | 164
percent change | -9.32 (1.362) | -8.53 (1.146)
Statistical Analysis 1: Comparison: CNM-Au8 vs Matching Placebo; Test type: Superiority; p = 0.6570, Mixed Models Analysis; Covariates include baseline use of edaravone and riluzole, months since symptom onset, and pre-baseline ALSFRS-R slope; Mean Difference (Net) = -0.78, 95% CI 2-sided [-4.25 to 2.68], Standard Error of Mean 1.766 — CNM-Au8 24-week change from baseline relative to placebo 24-week change from baseline

4. Secondary Outcome: Muscle Strength
Description: Change in muscle strength as measured isometrically using hand-held dynamometry (HHD).
Time Frame: Baseline to 24 Weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | CNM-Au8 | Matching Placebo
Number analyzed (Participants) | 120 | 164
percent change | -27.54 (2.647) | -24.44 (2.260)
Statistical Analysis 1: Comparison: CNM-Au8 vs Matching Placebo; Test type: Superiority; p = 0.3621, Mixed Models Analysis; Covariates include baseline use of edaravone and riluzole, months since symptom onset, and pre-baseline ALSFRS-R slope; Mean Difference (Net) = -3.10, 95% CI 2-sided [-9.78 to 3.58], Standard Error of Mean 3.403 — CNM-Au8 24-week change from baseline relative to placebo 24-week change from baseline

5. Secondary Outcome: Number of Participants That Experienced Death or Death Equivalent
Description: The number of participants who died or met the criterion for a death equivalent from the date of their baseline visit to the end of the Week 24visit window (generally 175 days after baseline). The death equivalent criterion is use of permanent assisted ventilation (PAV) for more than 22hours per day for more than 7 days in a row.
Time Frame: 24 Weeks
Population: Outcome measure data was analyzed using the Full Analysis Set (FAS), which includes shared placebo from other regimens.
Measure: Count of Participants; unit: Participants
Arm/Group | CNM-Au8 | Matching Placebo
Number analyzed (Participants) | 120 | 164
Participants | 3 | 5
Statistical Analysis 1: Comparison: CNM-Au8 vs Matching Placebo; Test type: Superiority; p = 0.7398, Log Rank

ADVERSE EVENTS:
Time Frame: Up to 35 weeks after participant signed Master Protocol consent.
Arm/Group | CNM-Au8 | Matching Placebo
All-Cause Mortality (participants affected / at risk) | 4/120 | 1/41
Serious Adverse Events (participants affected / at risk) | 16/120 | 7/41
Other Adverse Events (participants affected / at risk) | 110/120 | 38/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CNM-Au8 (N=120) | Matching Placebo (N=41)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Implant site cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Amyotrophic lateral sclerosis (Nervous system disorders) | 2 (2) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post-traumatic pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0)
Complication associated with device (Gastrointestinal disorders) | 1 (1) | 0 (0)
Failure to thrive (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CNM-Au8 (N=120) | Matching Placebo (N=41)
Muscular weakness (Nervous system disorders) | 24 (39) | 12 (17)
Headache (Nervous system disorders) | 17 (26) | 4 (6)
Neuromyopathy (Nervous system disorders) | 14 (21) | 6 (7)
Dysarthria (Nervous system disorders) | 15 (16) | 2 (2)
Tension headache (Nervous system disorders) | 7 (10) | 4 (4)
Amyotrophic lateral sclerosis (Nervous system disorders) | 6 (8) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 23 (33) | 4 (5)
Nausea (Gastrointestinal disorders) | 17 (21) | 6 (8)
Constipation (Gastrointestinal disorders) | 17 (19) | 3 (4)
Dysphagia (Gastrointestinal disorders) | 10 (10) | 5 (6)
Vomiting (Gastrointestinal disorders) | 6 (9) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 26 (44) | 13 (17)
Skin laceration (Injury, poisoning and procedural complications) | 6 (7) | 2 (2)
Post-traumatic pain (Injury, poisoning and procedural complications) | 3 (3) | 3 (3)
Fatigue (General disorders) | 13 (17) | 9 (9)
Oedema peripheral (General disorders) | 7 (13) | 4 (4)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 13 (14) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 (12) | 3 (3)
Urinary tract infection (Infections and infestations) | 10 (13) | 0 (0)
Sinusitis (Infections and infestations) | 6 (6) | 0 (0)
COVID-19 (Infections and infestations) | 2 (2) | 3 (3)
Weight Decreased (Investigations) | 2 (2) | 5 (5)
Depression (Psychiatric disorders) | 3 (3) | 4 (4)
Pruritus (Skin and subcutaneous tissue disorders) | 6 (8) | 0 (0)
Decreased Appetite (Metabolism and nutrition disorders) | 5 (5) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2021-11-22): https://cdn.clinicaltrials.gov/large-docs/45/NCT04414345/Prot_000.pdf
  • Statistical Analysis Plan (2022-07-22): https://cdn.clinicaltrials.gov/large-docs/45/NCT04414345/SAP_003.pdf